CLINICAL TRIAL: NCT06139978
Title: Is Size of Cisterna Magna Related to the Fetal Gender and Gestational Age
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alaa Gamal Abd El-Naser, Principal Investigator, Assiut University
Other Study IDs: CM.sex & age
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Size of Cisterna Magna; Gestational Age and Gender Conditions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women in male fetus: Mesurment size of cisterna magna and ather fetal biometric using 2D US
  Interventions: Behavioral: ultrasound observation
- Pregnant women in female fetus: Mesurment size of cisterna magna and ather fetal biometric using 2D US
  Interventions: Behavioral: ultrasound observation

INTERVENTIONS:
Behavioral: ultrasound observation — The relationship between the anteroposterior diameter of the CM and the gestational age and gender

SUMMARY:
The cisterna magna (CM) is a large subarachnoid cerebrospinal space that lies between the caudal aspect ofthe cerebellum and the medulla oblongata, drainingthe fourth ventricle . The evaluation of the fetal cisterna magna is animportant part of obstetric ultrasound which targetsdetection of prenatal malformation of the fetal centralnervous system (CNS).Therefore, measuring the size ofthe cisterna magna has important clinical significancefor diagnosing fetal nervous system abnormalities.

Studies about the relationship between the anteroposterior diameter of the CM and the gestational age (GA) are still controversial. Some articles havepointed out that there was a good correlationbetween the diameter of the CM and GA

DETAILED DESCRIPTION:
Prospective study that will include pregnant women who are between 20 weeks 0 days and 39 weeks 6 days of gestation. As in cross sectional study each fetus is considered only once. with use of magnetic resonance ultrasonography.( ultrasonography is a noninvasive imaging test uses high-frequency sound waves to create real-time pictures or video of internal organs or other soft tissues)

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are between 20 weeks 0 days and 39 weeks 6 days of gestation.
* Singleton pregnancy.

Exclusion Criteria:

.gestational age can not be confirmed.

* Fetal malformations or intrauterine growthretardation
* Women with chronic diseases.
* bodymass index >30

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Prospective study that will include pregnant women who are between 20 weeks 0 days and 39 weeks 6 days of gestation. As in cross sectional study each fetus is considered only once. with use of magnetic resonance ultrasonography.( ultrasonography is a noninvasive imaging test uses high-frequency sound waves to create real-time pictures or video of internal organs or other soft tissues).
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Correlation of cisterna magna size to the gender and gestational age | 48 months
  Mesurment of anteroposterior diameter of cisterna magna by centimeters using 2D US

CONTACTS AND LOCATIONS:
Overall Officials: Elwany D Elsenousy, professor, Study Chair — Assiut medical school
Locations (1):
- Assiut Medical School, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] McMillan JJ, Williams B. Aqueduct stenosis. Case review and discussion. J Neurol Neurosurg Psychiatry. 1977 Jun;40(6):521-32. doi: 10.1136/jnnp.40.6.521. PMID 302852
- [Result] D'Antonio F, Khalil A, Garel C, Pilu G, Rizzo G, Lerman-Sagie T, Bhide A, Thilaganathan B, Manzoli L, Papageorghiou AT. Systematic review and meta-analysis of isolated posterior fossa malformations on prenatal ultrasound imaging (part 1): nomenclature, diagnostic accuracy and associated anomalies. Ultrasound Obstet Gynecol. 2016 Jun;47(6):690-7. doi: 10.1002/uog.14900. Epub 2016 May 10. PMID 25970099
- [Result] Volpe P, Contro E, De Musso F, Ghi T, Farina A, Tempesta A, Volpe G, Rizzo N, Pilu G. Brainstem-vermis and brainstem-tentorium angles allow accurate categorization of fetal upward rotation of cerebellar vermis. Ultrasound Obstet Gynecol. 2012 Jun;39(6):632-5. doi: 10.1002/uog.11101. Epub 2012 May 14. PMID 22253138
- [Result] Araujo Junior E, Passos AP, Bruns RF, Nardozza LM, Moron AF. Reference range of fetal cisterna magna volume by three-dimensional ultrasonography using the VOCAL method. J Matern Fetal Neonatal Med. 2014 Jul;27(10):1023-8. doi: 10.3109/14767058.2013.847419. Epub 2013 Oct 22. PMID 24063432
- [Result] Araujo Junior E, Martins WP, Rolo LC, Pires CR, Zanforlin Filho SM. Normative data for fetal cisterna magna length measurement between 18 and 24 weeks of pregnancy. Childs Nerv Syst. 2014 Jan;30(1):9-12. doi: 10.1007/s00381-013-2298-y. PMID 24122018